CLINICAL TRIAL: NCT02137642
Title: A Single-center, Placebo-controlled, Double-blind, Study to Evaluate the Effects of RM-131 on Colonic Motor Functions in Patients With Chronic Constipation
Brief Title: Study to Evaluate the Effects of RM-131 in Patients With Chronic Constipation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Motus Therapeutics, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM-131-008
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Constipation
Keywords: constipation
MeSH Terms: conditions — Constipation | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RM-131 (Active Comparator)
  Interventions: Drug: RM-131
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RM-131 — Double blind RM-131 (100 ug) will be delivered once by injection during study procedure.
  Other Names: relamorelin
  Arms: RM-131
Drug: Placebo — Double blind placebo will be delivered once by injection during study procedure.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and tolerability as well as the effects of RM-131 on colonic motor and sensory effects in patients with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent prior to any study procedures, and be willing and able to comply with study procedures.
2. Subjects with chronic IDIOPATHIC constipation, including experiencing constipation for 12 or more weeks in the preceding 12 months. Chronic constipation is to be defined by the Rome III criteria for Functional Constipation
3. Stable concomitant medications defined as no changes in regimen for at least 2 weeks prior to the study period.
4. Body mass index of 18-40 kg/m2
5. Female patients must have negative urine pregnancy tests and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. Female patients unable to bear children must have this documented in their medical history. (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).

Exclusion Criteria:

1. Unable or unwilling to provide informed consent or to comply with study procedures
2. Diagnosis of secondary constipation e.g. underlying general neurological disease such as Parkinsonism, multiple sclerosis, diseases associated with peripheral neuropathy, iatrogenic constipation
3. Structural or metabolic diseases that affect the GI system NOTE: Patients with clinical suspicion of upper or lower GI obstruction must have been evaluated per standard of care and obstruction ruled out before screening
4. Unable to withdraw the following medications 48 hours prior to the colon study day and throughout the study:

   * Medications that alter GI transit including laxatives, magnesium and aluminum containing antacids, prokinetics, erythromycin, narcotics, aspirin, anti-cholinergics, tricyclic antidepressants, SNRI and newer antidepressants. With the exception of GoLYTELY which will be taken the evening prior to colon study day. 4- Selective serotonin reuptake inhibitor (SSRI) antidepressants are permissible at low, stable doses. All medications shall be reviewed and dis/approved by the principal investigator on a case by case basis.
   * Analgesic drugs including opiates, NSAIDs and COX-2 inhibitors
   * GABAnergic agents
   * Benzodiazepines NOTE: stable doses of thyroid replacement, estrogen replacement and birth control (but with adequate backup contraception as drug-interactions with birth control have not been conducted) are permissible.
   * Drugs with a low therapeutic index, such as warfarin, digoxin, anti-seizure medications
5. History of recent surgery (within 60 days of screening)
6. Acute or chronic illness or history of illness, which in the opinion of the Investigator, could pose a threat or harm to the patient or obscure interpretation of laboratory test results or interpretation of study data such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes, etc.
7. Any clinically significant abnormalities on physical examination or laboratory abnormalities identified in the medical record, as determined by the Investigator
8. Acute GI illness within 48 hours of initiation of the colonic study day
9. Females who are pregnant or breastfeeding
10. History of alcohol or substance abuse; Alcohol use 2 days before colonic study day
11. Participation in a clinical study involving an investigational medication within the 30 days prior to dosing in the present study
12. Any other reason, which in the opinion of the Investigator, would confound proper interpretation of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Effect of RM-131 on postprandial high amplitude propagated contractions (HAPC) per hour | Measured during the 2 hour study procedure
  Change from baseline HAPC

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Rochester, Rochester, Minnesota, United States